CLINICAL TRIAL: NCT05490693
Title: The Effect of Virtual Reality Glasses Used During Burn Dressing in Children on Pain, Anxiety and Fear
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, ümmühan kılıç, Principal Investigator, Ondokuz Mayıs University
Other Study IDs: OMU
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Randomized
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Experimental group — Experimental group: 26 control group group: 26
  Other Names: control group

SUMMARY:
This work; It was planned as a randomized controlled study to determine the effect of watching cartoons with virtual reality glasses during burn dressing of children aged 5-10 years who applied to the Training and Research Hospital Burn Unit Polyclinic on the feeling of pain, anxiety and fear in children.

DETAILED DESCRIPTION:
The study will be applied to children in the 5-10 group who will undergo burn dressing. During the dressing, children will be watched cartoons with virtual reality glasses and pain, anxiety and fear will be looked at before and after the dressing. The children in the control group will be given routine applications of the clinic.

ELIGIBILITY:
Inclusion Criteria:

* The child and family agree to participate in the research,
* The child does not have a disease that causes chronic pain,
* The child is between the ages of 5-10,
* 1st and 2nd degree burns of less than 10% of the body surface area of the child,
* Local burn, no facial burn
* The child has no mental or neurological disability
* Failure to intervene in the child with general anesthesia
* The child has no eye problems

Exclusion Criteria:

* Child and family refusal to participate in the study
* 3rd and 4th degree burns of more than 10% of the body surface area of the child,
* The child is less than 5 years old and over 10 years old
* The child has a mental or neurological disability
* Intervention of the child with general anesthesia
* The child has an eye problem

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In order to determine the number of samples, power analysis was performed using the G*power program. The effect size coefficient was calculated by using the Newcastle satisfaction scale averages in source 1 (thesis), and the effect size = 0.76, and it was decided to recruit at least 26 people in each group in order to obtain 80% power at the ɑ=0.05 level, a total of 52 people in the two groups.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
pain, anxiety, fear scores, | July 2022-October 2022
  We will evaluate the pain, anxiety, fear score with the Wong Baker Pain Scale before and after dressing in the trial and control group.reality glasses compared to the control group.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Omü, Samsun, İlkadım
  - 19May University, Samsun